CLINICAL TRIAL: NCT02226393
Title: Evaluating Effectiveness of Dyadic Prolonged Exposure Treatment on 2-4 Years Old vs. Toddler-parent Focused Treatment
Brief Title: Evaluating Effectiveness of Dyadic Prolonged Exposure on 2-4 Years Old vs. Toddler-parent Focused Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment
Sponsor: Association for Children at Risk (Other)
Collaborators: Geha Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC147804ctil
Record Dates: First submitted 2014-07-29; First posted 2014-08-27 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Post-Traumatic Stress Disorder in Children
Keywords: Toddlers; Preschoolers; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prolonged exposure (Experimental): See intervention description
  Interventions: Behavioral: Prolonged exposure
- Child-parent Play Therapy (Active Comparator): see intervention description
  Interventions: Behavioral: Child-parent Play Therapy

INTERVENTIONS:
Behavioral: Prolonged exposure — The PE treatment includes 12-15 60 minutes' sessions. The 2 main components of the treatment are psychoeducation about common reactions to trauma and in-vivo exposures (gradual exposure to trauma related situations and objects) and repeated recounting of the traumatic memory, Trauma memory recounting and in-vivo exposures are conducted during several successive sessions so the child learns that the exposures themselves pose no real harm to him, indicating that when one confronts what one is afraid of it becomes easier to manage.
  Arms: Prolonged exposure
Behavioral: Child-parent Play Therapy — Is consisted of 12-15 weekly 60 minute sessions of parent-child centered therapy it focus on establishing a trusting, empowering, and validating therapeutic relationship. Participants are allowed to choose when, how, and whether or not to address their trauma memory. Therapists provide active listening, empathy,and encouragement to talk about feelings and express belief in the participants ability to cope. In sessions 4 and 8, participants are asked how they feel about their trauma. With this exception, participants direct the sessions.
  Arms: Child-parent Play Therapy

SUMMARY:
Traumatic events have potentially debilitating long-lasting effects on the child's normal development and, therefore, should be effectively treated. Prolonged Exposure (PE) therapy has been found to be effective in reducing posttraumatic stress disorder symptoms in adults and in adolescents. It has not yet been tested in toddlers.

The purpose of this study is to examine the treatment efficacy of 2 methods of treatment for toddlers with PTSD and their parents. A randomized control trial could examine the efficacy of PE versus dyadic play therapy (TP-CT). Exploration of these questions under more rigorous conditions would help broaden our knowledge about developmentally sensitive treatment tools for this age group.

Our research hypotheses are:

1. PE would more effective than TP-CT in reducing post-traumatic symptoms in toddlers.
2. PE would more effective than TP-CT in reducing post-traumatic symptoms of the toddlers' parents.
3. These results will be preserved in a follow-up of 3-6 months post treatment. Following psychiatric assessment, 100 toddlers will be randomly assigned to PE and TP-CT (50 participants in each group).

DETAILED DESCRIPTION:
Beyond what was detailed in the previous section of the brief summary, it should be noted that the toddlers will be assessed and treated at least 1 month post-trauma and at least 1 month after discharge from hospital in order to avoid acute reaction either to the traumatic event or to the medical procedures during their hospitalization and adjustment problems.

ELIGIBILITY:
Inclusion Criteria:

1. Hebrew speaking toddlers with PTSD related to traumatic experience that occured at least 1 month prior to the study enrollment
2. Toddlers whose parents are living together

Exclusion Criteria:

1. Toddlers which are still dealing with an active life threatening illness and are hence going through medical procedures.
2. Toddlers with intelectual developmental disorder
3. Toddlers with an active psychosis
4. Toddlers with blindness or deafness
5. Toddlers who are currently taking psychotropic medication
6. Toddlers and parents that receive psycotherapy outside of the study for their PTSD symptoms
7. Toddlers diagnozed with autism spectrum disorder
8. Toddlers who were exposed to domestic or sexual violence

Ages: 18 Months to 66 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2014-10; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in post traumatic symptoms: clinical assessment and Young child ptsd checklist (YCPC, Scheeringa & Haslett, 2010). | Parents' pre-treatment, post treatment and follow-up 3,6,12 months post treatment
  Change from baseline in post traumatic symptoms will be assessed using the Classification of Mental Health and Developmental Disorders of Infancy and Early Childhood) and the Young Child PTSD Checklist (YCPC, Scheeringa & Haslett, 2010). The YCPC assesses probable diagnosis formed the basis for the new DSM-5 disorder for posttraumatic stress disorder for children 6 years and younger.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | Parents' pre-treatment, post treatment (after 12-15 sessions) and follow-up 3-6 months post treatment
  A self-report questionnaire for depression among adults
The Posttraumatic Stress Symptom Scale-Self report (PSS-SR; Foa, Riggs, Dancu & Rothbaum, 1993) | Parents' pre-treatment, during treatment (every 2 sessions), post treatment (after 12-15 sessions) and follow-up 3-6 months post treatment
  A self report questionnaire for the assessment of PTSD symptoms among adults
Posttraumatic Stress Cognitions Inventory (PTCI) | Parents' pre-treatment, post treatment (after 12-15 sessions) and follow-up 3-6 months post treatment
  A self report questionnaire assessing post traumatic beliefs in adults
Parenting Sense of Competence Scale )PSOC; Gibaud -Wallstton & Wandersman, 1978) | Parents' pre-treatment, post treatment (after 12-15 sessions) and follow-up 3-6 months post treatment
  The Parenting Sense of Competency Scale (PSOC) was developed by Gibaud-Wallston as part of her PhD dissertation and presented at the American Psychological Association by Gibaud-Wallston and Wandersman in 1978. The PSOC is a 17 item scale, with 2 subscales. Each item is rated on a 6 point Likert scale anchored by 1 = "Strongly Disagree" and 6 = "Strongly Agree".

CONTACTS AND LOCATIONS:
Overall Officials: Orit Krispin, Phd, Principal Investigator — Schneider Children's Medical Center, Israel; Lilach Rachamim, Phd, Study Director
Locations (2):
- Israel (2):
  - Rabin medical center, Petah Tikva
  - Association for Children at Risk's Cohen Harris Resilience Center, Tel Aviv